CLINICAL TRIAL: NCT06089785
Title: Evaluation of Splenic Stiffness in Liver Cell Failure Patients:Role of Elastography
Brief Title: Elastography in Liver Cell Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Omnia Saad Desoky Mohamed (Other)
Responsible Party: Sponsor-Investigator, Omnia Saad Desoky Mohamed, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: elastography in liver failure
Record Dates: First submitted 2023-09-29; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Liver Cell Damage
MeSH Terms: interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Samples not dependent on DNA of the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with liver cell failure: patients with liver cell failure and any complications
  Interventions: Device: elastography

INTERVENTIONS:
Device: elastography — evaluation of degree of spleen stiffness in liver cell failure patient by elastography.

SUMMARY:
1. evaluation of degree of spleen stiffness in liver cell failure patient by elastography.
2. correlation of degree of spleen stiffness and patient outcome

DETAILED DESCRIPTION:
Portal hypertension (PH) is a major complication of liver cirrhosis, as it predisposes to the development of serious clinical manifestations such as ascites, hepatic encephalopathy and variceal bleeding, aggravating the prognosis of patients.

Liver biopsy and hepatic venous pressure gradient (HVPG) measurements are the current gold standard procedures for determining fibrosis severity and diagnosing PH, respectively; however, both are invasive, limiting their use in clinical practice and larger trials of novel agents. Alternatively, many non-invasive methods have been proposed in order to substitute HVPG. Alterations in the biomechanical properties of the liver or spleen in patients with cirrhosis can be quantified by tissue elastography, which examines the elastic behavior of tissue after a force has been applied Among them, liver stiffness measurement (LSM) has been widely used, as it has been shown to correlate well with HVPG, though this relationship seems to weaken in values of HVPG higher than 12 mmHg, the threshold of serious complications development. Several studies supported the use of spleen stiffness measurement (SSM) instead of LSM, anticipating to a more adequate assessment of this advanced stage of PH. SS measured by ultrasound-based elastography showed good correlation with HVPG, detecting PH with a sensitivity and specificity of 0.88 and 0.92, respectively, and severe PH with a sensitivity and specificity of 0.92 and 0.79, respectively.The aim of this paper is to critically appraise and summarize the literature about the role of SSM as a predictive tool of liver decompensation and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age above 18 years. 2-patients with liver cell failure (hepatic encephalopathy, hematemesis, ascites, hepatocellular carcinoma) 3- patient height , Weight

Exclusion Criteria:

* 1- patients who refuse to contribute in this study. 2- Age below 18 years. 3-pregnancy and breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: any patient has any clinical picture for liver cell failure
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of splenic stiffness in liver cell failure patients: role of elastography | 4 years
  1. evaluation of degree of spleen stiffness in liver cell failure patient by elastography.
  2. correlation of degree of spleen stiffness and patient outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Result] Reiberger T. The Value of Liver and Spleen Stiffness for Evaluation of Portal Hypertension in Compensated Cirrhosis. Hepatol Commun. 2022 May;6(5):950-964. doi: 10.1002/hep4.1855. Epub 2021 Dec 14. PMID 34904404
- [Result] Yiyi M, Xiaoqin Q, Lei Z. Spleen Stiffness on Magnetic Resonance Elastography for the Detection of Portal Hypertension: A Systematic Review and Meta-Analysis. Iran J Public Health. 2022 Sep;51(9):1925-1935. doi: 10.18502/ijph.v51i9.10548. PMID 36743372